CLINICAL TRIAL: NCT00005984
Title: Autologous Marrow Transplantation for Chronic Myelogenous Leukemia Using Stem Cells Obtained After In Vivo Cyclophosphamide/G-CSF Priming
Brief Title: Cyclophosphamide and Filgrastim Followed By SCT in Patients With Chronic or Accelerated Phase Myelogenous Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated as principal investigator [PI] left the university.
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Catherine Verfaille, MD, Masonic Cancer Center, University of Minnesota
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1996LS183; UMN-MT-1996-11 (Other: Blood and Marrow Transplantation Program)
Record Dates: First submitted 2000-07-05; First posted 2003-01-27 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-09

CONDITIONS: Leukemia
Keywords: chronic phase myelogenous leukemia; accelerated phase myelogenous leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Chronic-Phase | interventions — Cyclophosphamide; Filgrastim; Interferon-alpha; Peripheral Blood Stem Cell Transplantation; Bone Marrow Transplantation; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients with CML (Experimental): Patients treated for chronic accelerated phase and/or chronic myelogenous leukemia (CML)
  Interventions: Drug: cyclophosphamide; Drug: filgrastim; Drug: recombinant interferon alfa; Procedure: peripheral blood stem cell transplantation; Procedure: radiation therapy

INTERVENTIONS:
Drug: cyclophosphamide — intravenously over 2 hours on day 1 and on days -7 and -6
  Other Names: Endoxan; Cytoxan
Drug: filgrastim — filgrastim (G-CSF) daily subcutaneously (SQ) starting on day 5 and continuing until completion of leukapheresis. Patients also receive G-CSF IV starting on day 0 and continuing until blood counts recover
  Other Names: NEUPOGEN®
Drug: recombinant interferon alfa — Beginning on Day 1, subcutaneous (SQ) daily administration in the absence of unacceptable toxicity or disease progression
  Other Names: INTRON® A
Procedure: peripheral blood stem cell transplantation — Patients receive the PBSC transplantation on day 0.
  Other Names: bone marrow transplant
Procedure: radiation therapy — total body irradiation twice a day on days -4 through -1
  Other Names: irradiation

SUMMARY:
RATIONALE: Giving colony-stimulating factors, such as G-CSF, and cyclophosphamide helps stem cells move from the patient's bone marrow to the blood so they can be collected and stored. Chemotherapy and radiation therapy is then given to prepare the bone marrow for the stem cell transplant. The stem cells are returned to the patient to replace the blood-forming cells that were destroyed by the chemotherapy and radiation therapy.

PURPOSE: This phase II trial is studying how well cyclophosphamide plus filgrastim followed by stem cell transplant works in treating patients with chronic phase or accelerated phase chronic myelogenous leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess the clinical outcomes, survival, and morbidity of patients with chronic or accelerated phase chronic myelogenous leukemia when treated with cyclophosphamide and filgrastim (G-CSF) followed by autologous peripheral blood stem cell transplantation.
* Determine whether priming with cyclophosphamide and filgrastim (G-CSF) increases the fraction of benign Philadelphia chromosome negative hematopoietic progenitors in peripheral blood stem cells (PBSC) and reduces the incidence of persistent or recurrent leukemia after autologous transplantation with mobilized PBSC in these patients.

OUTLINE: Patients receive priming therapy consisting of cyclophosphamide IV over 2 hours on day 1 and filgrastim (G-CSF) daily subcutaneously (SQ) starting on day 5 and continuing until completion of leukapheresis. Peripheral blood stem cells (PBSC) are collected between days 14-21.

Patients then receive preparative therapy for transplant consisting of cyclophosphamide IV over 2 hours on days -7 and -6 and total body irradiation twice a day on days -4 through -1. Patients receive the PBSC transplantation on day 0. Patients also receive G-CSF IV starting on day 0 and continuing until blood counts recover. Patients then receive interferon alfa SQ daily in the absence of unacceptable toxicity or disease progression.

Patients are followed at 3 weeks; then at 3, 6, 9, 12, and 18 months; and then annually for 5 years.

PROJECTED ACCRUAL: Not specified

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed chronic or accelerated phase chronic myelogenous leukemia (CML)

  * Philadelphia chromosome positive OR
  * BCR/ABL rearrangement
* Ineligible or refused to participate in ongoing allogeneic marrow donor transplant protocols
* 70 and under
* Performance status:

  * Age 65-70 years:
  * Karnofsky 80-100%
  * Under 65 years:
  * Karnofsky 90-100%
* Renal:

  * Age 65-70 years:
  * Creatinine clearance greater than 60 mL/min (if creatinine at least 1.5 mg/dL)
  * Under 65 years:
  * Not specified
* Cardiovascular:

  * Age 65-70 years:
  * LVEF at least 45%
* Pulmonary:

  * Age 65-70 years:
  * If history of smoking or respiratory symptoms, spirometry and DLCO must be greater then 50% of predicted
* Normal organ function (excluding bone marrow)

Exclusion Criteria:

* Blast crisis or post blast crisis
* Severe fibrosis defined by bilateral trephine biopsies
* Splenomegaly (below umbilicus) that does not respond to chemotherapy and/or radiotherapy

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2000-08; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Time to hemopoietic recovery after transplantation
Detection of the Philadelphia chromosome or the BCR/ABL gene abnormality in post-transplantation marrow samples

SECONDARY OUTCOMES:
Time to initial hospital discharge
Peritransplantation toxicity
Quality of life at various time points
Cause of death

CONTACTS AND LOCATIONS:
Overall Officials: Catherine M. Verfaillie, MD, Study Chair — Masonic Cancer Center, University of Minnesota
Locations (1):
- University of Minnesota Cancer Center, Minneapolis, Minnesota, United States